CLINICAL TRIAL: NCT02518321
Title: Can Technology-Assisted Toilets Improve Hygiene and Independence in Geriatric Rehabilitation? A Cohort Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: University of Ottawa (Other); Bruyère Academic Medical Organization (Unknown); TOTO USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: M16-15-022
Record Dates: First submitted 2015-07-03; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Geriatric Rehabilitation
Keywords: Toileting; Technology-Assisted Toilets; Rehabilitation; Assistive Devices; Activities of Daily Living

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Toileting First (Experimental): This group will complete the standard toileting trial before the TAT toileting trial.
  Interventions: Device: Technology-Assisted Toileting
- TAT Toileting First (Experimental): This group will complete the TAT toileting trial before the standard toileting trial.
  Interventions: Device: Technology-Assisted Toileting

INTERVENTIONS:
Device: Technology-Assisted Toileting
  Other Names: bidet toilets; smart toilets; TOTO Washlet

SUMMARY:
Toileting is a private activity of daily living. Geriatric rehabilitation patients are often unable to toilet themselves independently, leading to embarrassment and loss of self-esteem. Relationships with their caregivers may also become strained. Furthermore, improper toileting hygiene can lead to skin irritation, breakdown and infection.

Technology-assisted toilets (TATs) clean and dry the anal and vaginal regions using a stream of water and a fan. They can therefore potentially eliminate the need for patients to be able to wipe themselves. TATs are operated using wall-mounted remote controls. This study will examine the potential benefits of TAT use in geriatric rehabilitation patients.

Forty patients aged ≥65 years referred for treatment of physical impairments to the Geriatric Rehabilitation Unit (GRU) of the Elisabeth Bruyère Hospital (EBH) will be recruited for this study. Participants will have a bowel movement on two occasions, once using toilet paper and once using the TAT. The Psychosocial Impact of Assistive Devices Scale (PIADS), a validated questionnaire, will be used to analyze participants' toileting experience. Participants will be visually evaluated for cleanliness before and after each testing session.

The investigators hypothesize that participants will report that, in comparison with use of a standard toilet, toileting using the TAT: 1) is easier to use, 2) improves psychological well-being and 3) is more effective at cleaning than regular wiping techniques.

ELIGIBILITY:
Inclusion Criteria:

1. over the age of 65
2. inpatients at the EBH GRU
3. can communicate effectively in English or French
4. are able to remain balanced while sitting on a toilet
5. are able to physically use the remote control
6. are able to wipe themselves, but they do not need to be able to wipe themselves effectively

Exclusion Criteria:

1. are cognitively unable to provide informed consent
2. are severely aphasic
3. are undergoing treatment that interferes with toileting
4. have any conditions that increase perineal sensitivity such as ulcers, wounds, or infections
5. require two people to assist them in transferring to and from the toilet
6. are under isolation precautions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Psychosocial Impact of Assistive Devices Scale (PIADS) | up to 12 weeks
  Scale used to assess participants' subjective feelings of adaptability, competence, and self-esteem
Cleanliness Scale | up to 12 weeks
  A new scale being piloted to measure cleanliness of the anal/genital regions

CONTACTS AND LOCATIONS:
Overall Officials: Hillel Finestone, MD, Principal Investigator — Bruyère Continuing Care, Bruyère Research Institute, Elisabeth Bruyère Hospital, University of Ottawa.